CLINICAL TRIAL: NCT03368885
Title: Evaluation of Integrating Selected MIYCN Interventions in Existing Polio Eradication Platform of Project Concern International (PCI) in UP
Brief Title: Evaluation of Integrating MIYCN Interventions in Existing CGPP of PCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FHI 360 (Other)
Collaborators: International Food Policy Research Institute (Other); Project Concern International India (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1101870
Record Dates: First submitted 2017-11-29; First posted 2017-12-11 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Polio
Keywords: MIYCN -Maternal Infant Young Child Nutrition; CGPP - Core Group Polio Project; A&T- Alive and Thrive; PCI- Project Concern International; UP- Uttar Pradesh; VHSNC -Village Health, Sanitation and Nutrition Committee; CMC- Community Mobilization Coordinator
MeSH Terms: conditions — Poliomyelitis | interventions — Infant Nutritional Physiological Phenomena; Capacity Building

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental area PCI (Experimental): In this arm, in addition to the standard care for Polio eradication program activities of CGPP project, the following interventions are added:
  Maternal dietary diversity; Diet diversity in complementary feeding; Exclusive breast feeding; Community mobilization; Capacity building; Convergence;Use of existing platforms VHSND; Strategic Use of Data
  Interventions: Other: Maternal dietary diversity; Other: Diet diversity in complementary feeding; Other: Exclusive Breast Feeding; Other: Community mobilization; Other: Capacity Building; Other: Use of existing platforms VHSND; Other: Strategic use of data
- Control area PCI (No Intervention): This arm will receive standard care with respect to Polio eradication program activities of CGPP such as awareness generation around Polio and routine immunization, hand washing and sanitation

INTERVENTIONS:
Other: Maternal dietary diversity — Counsel pregnant women for proper dietary intake and create awareness among family members and community to support her on maternal nutrition
  Arms: Experimental area PCI
Other: Diet diversity in complementary feeding — Counsel mothers of children of 6-23 months on diet diversity in complementary feeding by demonstration during home-visits and seek support from father and family members
  Arms: Experimental area PCI
Other: Exclusive Breast Feeding — Counselling on exclusive breast feeding among children under 6 months-Provide information to mothers of children of 3-6 months for exclusive breast feeding through home visits, and mothers meetings
  Arms: Experimental area PCI
Other: Community mobilization — Engagement of local/religious leader, husbands to support diet diversity for pregnant women and doctors and fathers to support diet diversity for complementary feeding
  Arms: Experimental area PCI
Other: Capacity Building — Capacity Building-Training of Community mobilization coordinator and mentoring for knowledge enhancement on nutrition for pregnant women and children below 2 years
  Arms: Experimental area PCI
Other: Use of existing platforms VHSND — Convergence- Strengthen Village Health Sanitation and Nutrition Day for creating awareness on diet diversity for maternal nutrition and complementary feeding
  Arms: Experimental area PCI
Other: Strategic use of data — Strategic use of data-Data analysis for concurrent monitoring,planning and decision making to improve the performance of CMCs
  Arms: Experimental area PCI

SUMMARY:
The study has two arms; both experimental and control areas will receive standard interventions given under polio eradication program of PCI. Participants in the experimental arm receive additional interventions on nutrition (improve diet diversity in pregnant women and children of 6-23 months) for exact 12 months. The study includes awareness generation (regarding nutrition) through community mobilization, counseling and capacity building of community mobilization.

DETAILED DESCRIPTION:
The experimental arm will receive the following interventions:

1. Interpersonal communication (IPC) to reach target women (Women in their 2nd or 3rd trimester of pregnancy and women with 6-23 months old child) to deliver messages on maternal nutrition package and complementary feeding through home visits made by Community Mobilization Coordinator (CMC).
2. Expanded community mobilization involving key influencers in family like husbands and mothers -in-law and community opinion leaders, religious leaders, Village Health Sanitation and Nutrition Committee (VHSNC) members. The aims are to improve awareness, shift norms and perceptions, engage husbands and local opinion leaders to promote healthy behaviour practices related to maternal nutrition and complementary feeding.
3. Strategic use of data to design a context-specific program and track the progress of the program with regards to impact on social norms and behaviors at household/community level and demonstrate the feasibility of integrating select MIYCN interventions in polio eradication platforms.
4. Convergence: The convergence will mainly focus on three Cs - maintain consistency, avoid conflict and enhance cooperation. This will aid in passing consistent MIYCN messages to the target community and ensure effective teamwork, collaboration and mutual support

ELIGIBILITY:
Inclusion Criteria:

For Community

* • Women aged 15-49 years

  * Willing and able to provide consent
  * Women in 2nd and 3rd trimester of pregnancy and / or
  * Women with children aged 6-23 months For CMC
  * Women aged 18+
  * Currently appointed a CMC in a selected HRA
  * Willing and able to provide consent

Exclusion Criteria:

* Women in first trimester of pregnancy
* Women whose index child (youngest child, between 6-23 months of age) is not her biological child
* Women whose index child is not currently living with the mother

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2590 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-12-24 (Actual); Study Completion 2018-12-24 (Actual)

PRIMARY OUTCOMES:
Dietary Diversity in Maternal Nutrition | 12 months
  Percentage of Women in their 2nd or 3rd trimester of pregnancy from targeted households who consumed food from at least 5 specific nutrient rich food groups out of 10 defined food groups.
Minimum Dietary Diversity in Complementary Feeding | 12 months
  Percentage of children 6-23 months of age from targeted households who receive foods from 4 or more food groups (separately for breastfed and non-breastfed children)

SECONDARY OUTCOMES:
Timely Introduction of Complementary Feeding | 12 months
  Percentage of children 6-23 months of age who were initiated with complementary feeding in their seventh month.

CONTACTS AND LOCATIONS:
Overall Officials: Preeti Das, MPS, Principal Investigator — FHI 360
Locations (1):
- FHI Solutions LLC, Alive & Thrive, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided